CLINICAL TRIAL: NCT06435429
Title: A Phase 3, Randomized, Open-label, Multicenter, Controlled Study to Evaluate the Efficacy and Safety of Zanidatamab in Combination With Physician's Choice Chemotherapy Compared to Trastuzumab in Combination With Physician's Choice Chemotherapy for the Treatment of Participants With Metastatic HER2-positive Breast Cancer Who Have Progressed on, or Are Intolerant to, Previous Trastuzumab Deruxtecan Treatment
Brief Title: A Study Comparing the Efficacy and Safety of Zanidatamab to Trastuzumab, Each in Combination With Physician's Choice Chemotherapy, for the Treatment of Participants With Metastatic HER2-positive Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JZP598-303; 2023-508960-31-00 (Other: EU CTR)
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Metastatic HER2-positive Breast Cancer
Keywords: Zanidatamab; Trastuzumab; Metastatic HER2-positive breast cancer
MeSH Terms: interventions — zanidatamab; Trastuzumab; eribulin; Vinorelbine; Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zanidatamab plus physician's choice of chemotherapy (Experimental): Participants with HER2-positive metastatic breast cancer (mBC) who have progressed on, or are intolerant to, previous T-DXd treatment will be randomized to receive intravenous infusion of zanidatamab plus physician's choice of chemotherapy (eribulin, or vinorelbine, or gemcitabine, or capecitabine).
  Interventions: Drug: Zanidatamab; Drug: Eribulin; Drug: Vinorelbine; Drug: Gemcitabine; Drug: Capecitabine
- Trastuzumab plus physician's choice of chemotherapy (Active Comparator): Participants with HER2-positive metastatic breast cancer (mBC) who have progressed on, or are intolerant to, previous T-DXd treatment will be randomized to receive intravenous infusion of trastuzumab plus physician's choice of chemotherapy (eribulin, or gemcitabine, or vinorelbine, or capecitabine).
  Interventions: Drug: Trastuzumab; Drug: Eribulin; Drug: Vinorelbine; Drug: Gemcitabine; Drug: Capecitabine

INTERVENTIONS:
Drug: Zanidatamab — Administered by intravenous infusion
  Arms: Zanidatamab plus physician's choice of chemotherapy
Drug: Trastuzumab — Administered by intravenous infusion
  Arms: Trastuzumab plus physician's choice of chemotherapy
Drug: Eribulin — Administered by intravenous infusion
Drug: Vinorelbine — Administered by intravenous infusion
Drug: Gemcitabine — Administered by intravenous infusion
Drug: Capecitabine — Given orally

SUMMARY:
The efficacy and safety of zanidatamab in combination with physician's choice of chemotherapy compared with trastuzumab in combination with physician's choice of chemotherapy will be evaluated for the treatment of participants with metastatic HER2-positive breast cancer who have progressed on, or are intolerant to, previous T-DXd treatment.

DETAILED DESCRIPTION:
Zanidatamab, as a monotherapy or in combination with other antineoplastic agents, has shown clinically meaningful efficacy against multiple HER2-positive advanced/metastatic tumors, including in patients with metastatic breast cancer (mBC). Zanidatamab may offer a viable treatment option for patients with metastatic HER2-positive breast cancer.

The primary objective of the study is to compare the efficacy of zanidatamab plus chemotherapy versus trastuzumab plus chemotherapy. The secondary objectives of the study will include further comparing the efficacy, safety and tolerability, patient-reported tolerability, and patient-reported physical functioning of zanidatamab plus chemotherapy versus trastuzumab plus chemotherapy. The pharmacokinetics and immunogenicity of zanidatamab in combination with chemotherapy will also be evaluated.

ELIGIBILITY:
Participants are eligible to be included in the study only if all of the following criteria apply:

1. Is 18 years of age or of the legal adult age per local standard at the time of signing the informed consent.
2. Has histologically confirmed HER2-positive breast cancer according to ASCO-CAP Guidelines as evaluated by a sponsor-designated central laboratory
3. Participants with unresectable or metastatic HER2 positive breast cancer who have progressed on, or are intolerant to, previous T-DXd treatment.
4. Must have received at least 2 lines of HER2-directed therapy for their metastatic disease.

   1. Prior HER2-targeted neo-adjuvant or adjuvant therapy that resulted in relapse within 6 months of the completion of therapy will be considered a line of treatment for metastatic disease.
   2. Based on the physician's choice, participants' eligibility, and institutional and local guidelines, participants may also have received post-T-DXd therapy, for example, a tucatinib-based regimen and/or T-DM1.
   3. Participants must not have received more than 4 lines of HER2-directed therapy in the metastatic setting.
5. Has measurable disease per RECIST version 1.1.
6. Is eligible to receive one of the chemotherapy options listed in the physician's choice of chemotherapy (eribulin, gemcitabine, vinorelbine, or capecitabine).
7. Participants with history of treated or clinically inactive CNS metastases are eligible as specified in the protocol.
8. Has a life expectancy of at least 6 months, in the opinion of the investigator.
9. Has adequate hematologic parameters as defined in the protocol.
10. Has adequate hepatic function as specified in the protocol.
11. Has creatinine clearance ≥ 50 mL/minute as calculated per local institutional guidelines.
12. Has LVEF ≥ 50% as determined by either echocardiogram or MUGA obtained within 4 weeks before the first dose of study intervention.
13. Has ECOG performance status of 0 or 1.
14. Participant agrees to the following based on sex assigned at birth.

    1. Male participants:

       Male participants are eligible to participate if they agree to the following during the study intervention period and for at least 7 months after the last dose of study intervention or the contraception period for the combination chemotherapy of choice per local guidance/standard practice:
       * Refrain from donating fresh unwashed semen.
       * Use contraception as follows as specified in the protocol
    2. Female participants:

       * A female participant is eligible to participate if she is not pregnant or breastfeeding, and one of the following conditions applies:

         * Is a women of nonchildbearing potential OR
         * Is a woman of childbearing potential (WOCBP) and using a contraceptive method that is highly effective (with a failure rate of < 1% per year), with low user dependency during the study intervention period and for at least 7 months after the last dose of study intervention.
       * A WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 3 days before the first dose of study intervention.
       * Additional requirements for pregnancy testing during and after study intervention are provided in the protocol.
       * The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
15. Is capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form and in the protocol.

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. Has clinically confirmed leptomeningeal disease, in the opinion of the investigator.
2. Has uncontrolled or significant cardiovascular disease.
3. Has toxicity related to prior cancer therapy that has not resolved to ≤ Grade 1, with exceptions as stated in the protocol.
4. Has uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.
5. Has an infection with HIV-1 or HIV-2, with the exception of participants with well-controlled HIV.
6. Has active hepatitis B or C infection.
7. Has an active SARS-CoV-2 infection. Participants with prior infection that has resolved per local institutions' requirements and screening guidance are eligible.
8. Has a history of life-threatening hypersensitivity to monoclonal antibodies or to recombinant proteins or excipients in the drug formulation of zanidatamab.
9. Is unable to receive trastuzumab treatment due to medical contraindications.
10. Has any serious underlying medical or psychiatric condition that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site.
11. Has any condition that would prevent treatment with the physician's choice of chemotherapy.
12. Has any issue or condition that in the opinion of the investigator would contraindicate the participant's participation in the study or confound the results of the study.

    Prior/Concomitant Therapy
13. Has a history of prior allogeneic bone marrow, stem cell, or solid organ transplantation.
14. The washout periods for prior anticancer therapies before randomization as specified in the protocol.
15. Has a history of trauma or major surgery within 4 weeks prior to randomization.

    Other Exclusions
16. Has a known hypersensitivity to any components of the study drugs, including chemotherapy.
17. Female participants who are breastfeeding or pregnant, and female and male participants planning a pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2028-04-28 (Estimated); Study Completion 2030-10-18 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) Per RECIST Version 1.1 As Assessed by Blinded Independent Central Review (BICR) | Until disease progression or death, up to approximately 44 months
  PFS is defined as the time in months from randomization to the date of first documented disease progression (as assessed by BICR according to RECIST v1.1) or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Until death, up to approximately 80 months
  OS is defined as the time in months from randomization to the date of death due to any cause.
Confirmed Objective Response Rate (ORR) Per RECIST Version 1.1, As Assessed by BICR | Until disease progression or death, up to approximately 44 months
  The BICR-assessed confirmed ORR is defined as the proportion of participants who had a best overall response of BICR-assessed Complete Response (CR) or Partial Response (PR) after randomization.
Duration of Response (DOR) Per RECIST Version 1.1, As Assessed by BICR | Until disease progression or death, up to approximately 44 months
  BICR-assessed DOR is defined as the time in months from the first objective response (CR or PR) that is subsequently confirmed to documented progressive disease (PD) as assessed by BICR per RECIST v1.1 or death from any cause.
PFS Per RECIST Version 1.1, As Assessed By Investigator | Until disease progression or death, up to approximately 44 months
  Investigator-assessed PFS is defined as the time in months from randomization to the date of first documented disease progression (as assessed by investigator according to RECIST v1.1) or death from any cause, whichever occurs first
Confirmed ORR Per RECIST Version 1.1, As Assessed By Investigator | Until disease progression or death, up to approximately 44 months
  The investigator-assessed confirmed ORR is defined as the proportion of participants who had a best overall response of investigator-assessed confirmed CR or PR after randomization.
DOR Per RECIST Version 1.1, As Assessed By Investigator | Until disease progression or death, up to approximately 44 months
  Investigator-assessed DOR is defined as the time in months from the first objective response (CR or PR) that is subsequently confirmed to documented PD as assessed by the investigator per RECIST v1.1 or death from any cause.
Number of Participants Reporting Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events As Graded by NCI CTCAE Version 5.0 | Up to approximately 44 months
Number of Participants With Dose Reductions | Up to approximately 44 months
Number of Participants Discontinuing Study Treatment Due to TEAEs | Up to approximately 44 months
Serum Concentrations of Zanidatamab | Up to approximately 44 months
Number of Participants Positive for Anti-drug Antibodies to Zanidatamab | Up to approximately 44 months
Proportion of All Treated Participants, As Treated, Reporting Symptomatic Adverse Events While On Treatment Based on Patient-reported Outcome-Common Terminology Criteria for AEs and European Organisation for Research and Treatment of Cancer Item Library | Up to approximately 44 months
Proportion of All Treated Participants, As Treated, Reporting Overall Side-effect Bother on the Functional Assessment of Chronic Illness Therapy General Physical Item 5 (FACIT-GP5) | Up to approximately 44 months
  The Functional Assessment of Chronic Illness Therapy (FACIT) GP5 Item score ranges from 0 (Not at all) to 4 (Very Much), where higher scores reflect greater bother from treatment side effects.
Proportion of Treated Participants, As Treated, With Maintained or Improved Physical Function While On Treatment Based On The Physical Functioning Subscale of the EORTC Quality of Life Questionnaire Core Module (EORTC QLQ-C30) | Up to approximately 44 months
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core Module Physical Functioning score ranges from 0 to 100, where higher scores reflect better functioning.

CONTACTS AND LOCATIONS:
Locations (166):
- United States (48):
  - Mayo Clinic Scottsdale - PPDS, Phoenix, Arizona
  - Arizona Oncology Tucson - Wilmot, Tucson, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - The Oncology Institute Of Hope And Innovation, Cerritos, California
  - Los Angeles Hematology Oncology Medical Group Glendale, Glendale, California
  - USC-Norris Comprehensive Cancer Center - Investigational Drug Service IDS, Los Angeles, California
  - UCSF at Mission Bay MB, San Francisco, California
  - University of Colorado-Cancer Center-PPDS, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Washington Cancer Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists Research South, Fort Myers, Florida
  - Mayo Clinic Jacksonville - PPDS, Jacksonville, Florida
  - Florida Cancer Specialists Research North, St. Petersburg, Florida
  - Florida Cancer Specialists Research East, West Palm Beach, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Minnesota Oncology Hematology, Coon Rapids, Minnesota
  - Mayo Clinic - PPDS, Rochester, Minnesota
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering, Long Island City, New York
  - Perlmutter Cancer Center 160 E 34th St, New York, New York
  - The Mount Sinai Hospital, New York, New York
  - Columbia University Medical Center 161 Fort Washington, New York, New York
  - Messino Cancer Center, Asheville, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - UNC Central Investigational Drug Services, Morrisville, North Carolina
  - Oncology Hematology Care (OHC), Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center 11100 Euclid Ave, Cleveland, Ohio
  - Abramson Cancer Center of The University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - U.T. MD Anderson Cancer Center, Investigational Pharmacy Services, Houston, Texas
  - Millennium Research and Clinical Development, Houston, Texas
  - Maryland Oncology Hematology Healing Way - USOR, Irving, Texas
  - Medical Oncology Hematology Consultants, Irving, Texas
  - Nexus Health, Irving, Texas
  - Sansum Clinic 540 W - USOR, Irving, Texas
  - Texas Oncology Gulf Coast, Irving, Texas
  - Texas Oncology West, Irving, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Sentara Health, Norfolk, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (6):
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - Box Hill Hospital, Melbourne, Victoria
  - Peninsula and South Eastern Haematology and Oncology Group, Mount Waverly, Victoria
  - HPS Pharmacies - Adelaide, Adelaide
  - The Kinghorn Cancer Centre, Mount Kuring-Gai
  - St John of God Hospital Subiaco, Subiaco
- Austria (4):
  - Medizinische Universitat Innsbruck, Innsbruck
  - Ordensklinikum Barmherzige Schwestern, Linz
  - Medizinische Universitat Wien, Vienna
  - Klinikum Wels-Grieskirchen GmbH - Abteilung für Innere Medizin IV, Wels
- Belgium (5):
  - Institute Jules Bordet, Anderlecht
  - UZ Antwerpen, Edegem
  - Grand Hôpital de Charleroi, Gilly
  - CHU UCL Namur - Site Sainte-Elisabeth, Namur
  - AZ Delta- Campus Rumbeke, Roeselare
- Brazil (12):
  - Hospital Nossa Senhora Da Conceição, Porto Alegre, Rio Grande do Sul
  - IEPE Unimed Sorocaba, Sorocaba, São Paulo
  - DASA Hospital Brasilia, Brasília
  - Centro Regional Integrado de Oncologia, Ceará
  - Catarina Pesquisa Clinica, Itajaí
  - Irmandade Da Santa Casa de Misericordia de Porto Alegre, Portalegre
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul PUCRS, Porto Alegre
  - Real Hospital Portugues de Beneficiencia Em Pernambuco, Recife
  - Nucleo de Oncologia Da Bahia, Salvador
  - Ceon Pesquisas Ltda, São Caetano do Sul
  - Hospital Beneficiencia Portuguesa, São Paulo
  - Onco Star Sp Oncologia LTDA, São Paulo
- Canada (5):
  - Jewish General Hospital, Montreal
  - The Ottawa Hospital Cancer Centre, Ottawa
  - CHU de Québec Université Laval Hôpital du Saint Sacrement, Québec
  - Sunnybrook Research Institute, Toronto
  - BC Cancer-Vancouver Center, Vancouver
- France (11):
  - Institut Bergonie, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Pharmacie Centre de Cancerologie de la Sarthe, Le Mans
  - Centre Oscar Lambret, Lille
  - AP HM Hopital de La Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - Pharmacie ICM Val d'Aurelle, Montpellier
  - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Oncopôle Claudius Regaud Pharmacie, Toulouse
  - Gustave Roussy, Villejuif
- Germany (5):
  - Helios Klinikum Berlin Buch GmbH Klinik für Gynäkologie und Geburtshilfe, Berlin
  - Marienhospital Bottrop gGmbH, Dortmund
  - Universitätsklinikum Carl Gustav Carus an der TU, Dresden
  - LMU Klinikum - Apotheke, München
  - Universitätsklinikum Ulm, Ulm
- Greece (4):
  - Aretaieio Hospital, Athens
  - Athens Medical Center, Athens
  - University General Hospital of Patras, Pátrai
  - European Interbalkan Medical Center, Thessaloniki
- Italy (11):
  - IRCCS Centro di Riferimento Oncologico di Aviano CRO, Aviano
  - Asst Papa Giovanni Xxiii, Bergamo
  - Azienda Ospedaliero Universitaria Di Bologna Policlinico S Orsola Malpighi Via Massarenti, Bologna
  - Ospedale San Raffaele S.r.l PPDS, Milan
  - Istituto Europeo di Oncologia, Milan
  - Azienda Ospedaliero Universitaria di Modena, Modena
  - Fondazione IRCCS San Gerardo dei Tintori, Monza
  - Istituto Oncologico Veneto - I.R.C.C.S., Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome
  - IRCCS Istituto Clinico Humanitas, Rozzano
- Japan (17):
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital, Chūōku
  - Osaka International Cancer Institute, Chūōku
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Saitama Medical University International Medical Center, Hidaka-shi
  - Tokai University Hospital, Isesaki-shi
  - Sagara Hospital, Kagoshima
  - Kyoto University Hospital, Kyoto
  - Aichi Cancer Center, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Okayama University Hospital, Okayama
  - National Hospital Organization Osaka National Hospital, Osaka
  - National Hospital Organization Hokkaido Cancer Center, Sapporo
  - Juntendo University Hospital, Tokyo
  - Showa University Hospital, Tokyo
  - Kanagawa Cancer Center, Yokohama
- Poland (6):
  - Białostockie Centrum Onkologii im. Marii Skłodowskiej-Curie w Białymstoku, Bialystok
  - Wojewódzki Szpital Specjalistyczny W Białej Podlaskiej, Biała Podlaska
  - Pratia MCM Kraków, Krakow
  - Pratia Poznan, Poznan
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy w Warszawie, Warsaw
- South Korea (8):
  - Soon Chun Hyang University Cheonan Hospital, Cheonan-si
  - Gachon University Gil Medical Center, Namdong-gu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (16):
  - Hospital Universitario A Coruña, A Coruña
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - ICO Badalona-H.U. Germans Trias i Pujol, Barcelona
  - Hospital General Universitario de Elche, Elche
  - Hospital Universitario Clinico San Cecilio, Granada
  - Hospital Beata Maria Ana, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo
- United Kingdom (8):
  - Royal United Hospital, Bath
  - Beatson West Of Scotland Cancer Centre, Glasgow
  - Leicester Royal Infirmary, Leicester
  - Guy's Hospital, London
  - Charring Cross Hospital, London
  - The Christie - PPDS, Manchester
  - Churchill Hospital, Oxford
  - New Cross Hospital, Wolverhampton

IPD SHARING:
Plan to Share IPD: No